CLINICAL TRIAL: NCT02643459
Title: Introduction of Soluble Urokinase Plasminogen Activating Receptor in Acute Care as a Prognostic Biomarker to Strengthen Risk Stratification of Acutely Admitted Patients
Brief Title: Risk Stratification in Acute Care: The Meaning of suPAR Measurement in Triage
Acronym: suPAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Martin Schultz, MD, P.h.D student, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HerlevH01
Record Dates: First submitted 2015-11-13; First posted 2015-12-31 (Estimated); Results first posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Triage; Risk Stratification With Biomarker
Keywords: Triage; Risk stratification; Acute care; suPAR

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional (No Intervention): no suPAR measurement. Standard care.
- suPAR (Experimental): suPAR measurement and education of doctors working in the Emergency department in the meaning of low or elevated levels of suPAR. Since suPAR is measured on all patients regardless of disease the investigators cannot define a single intervention. A possible intervention depends on the clinical situation.
  Interventions: Behavioral: suPAR measurement

INTERVENTIONS:
Behavioral: suPAR measurement — The biomarker suPAR will be measured on all patients included in the study. Before the study period the doctors will receive information on suPAR. We want to study if the information provided by suPAR is useful in emergency medicine. Interventions depends on the clinical issue, as suPAR is an unspecific marker of disease. Usually a elevated suPAR level could result in more investigation e.g. diagnostic procedures or follow up, while a low suPAR could result in faster discharge.
  Arms: suPAR

SUMMARY:
Will clinical outcome for patients be improved if triage in Acute wards and Emergency rooms is supplemented with a prognostic biomarker?

DETAILED DESCRIPTION:
In a health care system where the general population is growing, more patients are living with chronic conditions and the hospitals are reducing beds and length of stay, it is crucial to perform safe and fast risk stratification of patients presenting in the Emergency departments. Risk stratification is currently performed with a combination of measurement of the vital signs and assessment of the primary complaint. The aim of the current study is to assess whether the supplement of biomarkers can improve the risk stratification in regard to mortality, readmissions and improve overall patient flow in the Emergency departments. Soluble urokinase plasminogen activating receptor (suPAR) is the soluble form of urokinase-type plasminogen activator receptor (uPAR). uPAR is present on various immunological active cells, as well as endothelia and smooth muscle cells. It is believed that suPAR mirrors the inflammatory response in patients. Previous studies have shown a strong association with mortality and severity of disease in a broad variety of conditions (infection, hepatic-, renal-, cardiac- and lung disease) as well as a possible marker of disease development in the general population. These abilities indicate that suPAR although unspecific would be ideal to identify patients at high- and at low-risk. The aim is to target interventions and limited clinical focus where it is most beneficial. In unselected patients suPAR is one of the strongest prognostic biomarker available to date.

It is not known whether information on prognosis in the Emergency department can be used to prevent death, serious complications or reduce admissions and readmissions.

The purpose of the current study is to examine if introduction of the biomarker suPAR and education of doctors in the meaning of suPAR levels and association to disease, can reduce mortality, admissions and readmission in patients referred to the emergency rooms.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting acutely to the Acute ward/Emergency department and have blood samples done which include both Hemoglobin, C reactive protein and Creatinine within 6 hours of registration within the study period. The study is carried out in 2 Hospitals in the Capital of Denmark.

Exclusion Criteria:

* Patients presenting in Pediatric, Gynecological or Obstetric units. Patients not being examined with blood samples.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20000 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kasper K Iversen, MD, DMSci, Study Director — Department of Cardiology, Herlev Hospital
Locations (1):
- Herlev Hospital, Department of Cardiology, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schultz M, Rasmussen LJH, Hoi-Hansen T, Kjoller E, Jensen BN, Lind MN, Ravn L, Kallemose T, Lange T, Kober L, Rasmussen LS, Eugen-Olsen J, Iversen KK. Early Discharge from the Emergency Department Based on Soluble Urokinase Plasminogen Activator Receptor (suPAR) Levels: A TRIAGE III Substudy. Dis Markers. 2019 May 19;2019:3403549. doi: 10.1155/2019/3403549. eCollection 2019. PMID 31236143
- [Derived] Schultz M, Rasmussen LJH, Kallemose T, Kjoller E, Lind MN, Ravn L, Lange T, Kober L, Rasmussen LS, Eugen-Olsen J, Iversen K. Availability of suPAR in emergency departments may improve risk stratification: a secondary analysis of the TRIAGE III trial. Scand J Trauma Resusc Emerg Med. 2019 Apr 11;27(1):43. doi: 10.1186/s13049-019-0621-7. PMID 30975178
- [Derived] Schultz M, Rasmussen LJH, Andersen MH, Stefansson JS, Falkentoft AC, Alstrup M, Sando A, Holle SLK, Meyer J, Tornkvist PBS, Hoi-Hansen T, Kjoller E, Jensen BN, Lind M, Ravn L, Kallemose T, Lange T, Kober L, Rasmussen LS, Eugen-Olsen J, Iversen KK. Use of the prognostic biomarker suPAR in the emergency department improves risk stratification but has no effect on mortality: a cluster-randomized clinical trial (TRIAGE III). Scand J Trauma Resusc Emerg Med. 2018 Aug 28;26(1):69. doi: 10.1186/s13049-018-0539-5. PMID 30153859
- [Derived] Sando A, Schultz M, Eugen-Olsen J, Rasmussen LS, Kober L, Kjoller E, Jensen BN, Ravn L, Lange T, Iversen K. Introduction of a prognostic biomarker to strengthen risk stratification of acutely admitted patients: rationale and design of the TRIAGE III cluster randomized interventional trial. Scand J Trauma Resusc Emerg Med. 2016 Aug 5;24:100. doi: 10.1186/s13049-016-0290-8. PMID 27491822

RESULTS

PARTICIPANT FLOW:
Groups:
- suPAR: suPAR measurement and education of doctors working in the Emergency department in the meaning of low or elevated levels of suPAR.
Period: Overall Study
Arm/Group | Conventional | suPAR
Started | 7901 | 8900
Completed | 7901 | 8900
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional | suPAR | Total
Number analyzed (Participants) | 7901 | 8900 | 16801
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (20.7) | 60.4 (20.8) | 60.6 (20.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4175 | 4689 | 8864
  Male | 3726 | 4211 | 7937
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 7901 | 8900 | 16801
Region of Enrollment [Number; unit: participants]
  Denmark | 7901 | 8900 | 16801

OUTCOME MEASURES:

1. Primary Outcome: All Cause Mortality
Description: Time frame starts at the beginning of the index admission, defined as first admission in the study period. Patients will be followed using central registers.
Time Frame: 10 months after the inclusions period ends mortality data will be assessed
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional | suPAR
Number analyzed (Participants) | 7901 | 8900
Participants | 1126 | 1241

2. Secondary Outcome: All Cause Mortality
Description: Mortality within 30 days
Time Frame: 1 months after index admission mortality data will assessed
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional | suPAR
Number analyzed (Participants) | 7901 | 8900
Participants | 319 | 359

3. Secondary Outcome: Number of Discharges From the Emergency Room Within 24 Hours
Description: How many patients are discharged directly from the ED
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional | suPAR
Number analyzed (Participants) | 7901 | 8900
Participants | 3934 | 4352

4. Secondary Outcome: Number of Admissions to the Medical Ward
Description: Number of Participants with Admissions to the Medical War
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional | suPAR
Number analyzed (Participants) | 7901 | 8900
Participants | 3500 | 3738

5. Secondary Outcome: Number of Patients With an Admission to the Intensive Care Unit
Description: Number of Participants with transfer to the ICU
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional | suPAR
Number analyzed (Participants) | 7901 | 8900
Participants | 1027 | 1157

6. Secondary Outcome: Number of Patients With New Cancer Diagnosis in Control vs Intervention Groups
Time Frame: 10 months after inclusion period ends
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional | suPAR
Number analyzed (Participants) | 7901 | 8900
Participants | 687 | 917

7. Secondary Outcome: Length of Stay During Admission.
Description: Length of stay in days during the admission
Time Frame: 30 days
Measure: Mean (Standard Error); unit: Days
Arm/Group | Conventional | suPAR
Number analyzed (Participants) | 7901 | 8900
Days | 4.53 (8.7) | 4.39 (8.27)

8. Secondary Outcome: Number of Readmissions
Description: Patients will be followed using central registers. All new admissions within 90 days of the same patient is defined as readmissions.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Conventional | suPAR
Number analyzed (Participants) | 7901 | 8900
Participants | 687 | 917

ADVERSE EVENTS:
Time Frame: 1 year
Description: Data on all outcomes were collected from national registries.
Arm/Group | Conventional | suPAR
All-Cause Mortality (participants affected / at risk) | 1126/7901 | 1241/8900
Serious Adverse Events (participants affected / at risk) | 0/7901 | 0/8900
Other Adverse Events (participants affected / at risk) | 700/7901 | 777/8900
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional (N=7901) | suPAR (N=8900)
New cancer diagnosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 700 (700) | 777 (777)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/59/NCT02643459/Prot_SAP_000.pdf